CLINICAL TRIAL: NCT01133002
Title: National, Prospective, Observational, Cohort Study of Venous Thromboembolism (VTE) Management With the Low Molecular Weight Heparin, Enoxaparin, in the Outpatient Setting in Canada
Brief Title: Canadian Outpatient VTE Management Registry
Acronym: RECOVERY
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs study director, sanofi-aventis
Other Study IDs: ENOXA_L_02260
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Medical Prevention Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- VTE management registry: Patients receiving enoxaparin, with or without oral anticoagulation, within Day 0-10 after diagnosis of VTE

SUMMARY:
Primary Objective:

- To obtain prospective, clinical practice-based data on how symptomatic VTE is managed with low molecular weight heparin (LMWH) enoxaparin in Canadian outpatient settings.

Secondary Objective:

* To describe the demographic and clinical characteristics of patients with symptomatic VTE including characteristics of VTE, VTE risk factors and bleeding risk factors.
* To assess the frequency of patient characteristics that would necessitate adjustment in the dose or duration of enoxaparin therapy, e.g. high BMI, impaired creatinine clearance, advanced age, cancer-associated VTE.
* To assess the degree of adherence in clinical practice to Consensus Guidelines (ACCP/American College of chest Physician 2008) for the management of acute VTE, vis a vis:
* Appropriate dosing of enoxaparin
* Recommended duration of initial LMWH therapy
* Adequate overlap of LMWH with vitamin K antagonists (VKA)
* Recommended duration of longterm VKA
* Frequency of use of LMWH monotherapy to treat cancer-related VTE
* To access safety outcomes (including bleeding and recurrent VTE)
* To describe the utilization of resources due to bleeding and recurrent VTE during the treatment period.

ELIGIBILITY:
Inclusion criteria:

* Objectively confirmed VTE
* Initiation of enoxaparin treatment within Day 0-10 after diagnosis of VTE:
* Outpatients who will be treated with enoxaparin + VKA in combination are permitted to receive initial treatment other than enoxaparin for a maximum of 48 hours or 2 treatment doses preceding entry into the study
* Outpatients on enoxaparin monotherapy are permitted to receive up to 10 days of treatment other than enoxaparin preceding entry into the study.

Exclusion criteria:

- Medical or psychiatric disorders associated with altered cognition or mentation that precludes understanding of the informed consent process.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with objectively confirmed symptomatic VTE treated at approximately 15 outpatient clinics across Canada which use enoxaparin for the treatment of acute VTE.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Deep Venous Thrombosis (DVT) and/or Pulmonary Embolism (PE) and/or thrombosis at unusual sites | Day 180 or end of anticoagulant therapy whichever comes first
Number of patients prescribed twice daily (BID) vs. once daily (QD) enoxaparin | Day 180 or end of anticoagulant therapy whichever comes first
Proportion of patients who used short (5-7 days) vs. longer use (more than 7 days) durations of treatment with enoxaparin | Day 180 or end of anticoagulant therapy whichever comes first
Percentage of exnoxaparin prefilled syringes vs. multidose vials used during treatment | Day 180 or end of anticoagulant therapy whichever comes first

SECONDARY OUTCOMES:
Patient characteristics associated with different patterns of VTE management and enoxaparin use | Day 180 or end of anticoagulant therapy whichever comes first
  Analysis of patient characteristics associated with different patterns of VTE management and enoxaparin use, such as age, weight, creatinine clearance, co-morbid disease, VTE characteristics, concomitant use of other pharmacological and non-pharmacological treatment of the VTE, concomitant use of other non-VTE related therapies
Percentage of cases managed as recommended by Concensus Guidelines (ACCP 2008) | Day 180 or end of anticoagulant therapy whichever comes first
Incidence of bleeding events and episodes of recurrent VTE | Day 180 or end of anticoagulant therapy whichever comes first
To tabulate VTE-related resources utilized during the study period and compare resource utilization in patients treated vs not treated as per Concensus Guidelines (ACCP 2008) | Day 180 or end of anticoagulant therapy whichever comes first
  VTE-related resources utilized during the study period, including cost of VTE and its treatment (e.g. duration of hospital stay, drug costs, costs related to bleeding such as transfusions, costs of recurrent VTE) and compare resource utilization in patients treated vs. not treated as recommended by Concensus Guidelines (ACCP 2008)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada